CLINICAL TRIAL: NCT06868134
Title: The Effectiveness of Different Exercise Application Methods in Postmenopausal Women
Brief Title: Efficacy of Exercise Methods in Postmenopausal Women: a Clinical Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, dogukan kurc, Lecturer, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E-10840098-772.02-4975
Record Dates: First submitted 2025-03-05; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Post Menopausal Women

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (No Intervention): Participants in this group will not receive any intervention
- Supervised Exercise Group (Experimental): Participants in this group will receive a supervised progressive exercise program including stretching, strengthening, and aerobic exercises. The intervention will be performed 3 times per week with at least one rest day between sessions.
  Interventions: Behavioral: Supervised Progressive Exercise Program
- Web-Based Exercise Group (Experimental): Participants in this group will follow a progressive exercise program through the Physitrack web platform. At the beginning and at the end of the 8th week, participants will be assessed. A profile will be created for each participant by the researcher, and the individualized progressive exercise program will be assigned to their profiles. The intervention will be performed 3 times per week with at least one rest day between sessions.
  Interventions: Behavioral: Web-Based Exercise Group

INTERVENTIONS:
Behavioral: Web-Based Exercise Group — Participants will follow a structured progressive exercise program through the Physitrack web platform, including stretching, strengthening, and aerobic exercises. The program will be assigned to each participant's profile, and they will complete the exercises three times per week with at least one rest day between sessions. Assessments will be conducted at the beginning and at the end of the 8th week.
  Arms: Web-Based Exercise Group
Behavioral: Supervised Progressive Exercise Program — Participants in this group will receive a supervised progressive exercise program consisting of stretching, strengthening, and aerobic exercises. The intervention will be conducted three times per week with at least one rest day between sessions.
  Arms: Supervised Exercise Group

SUMMARY:
This study aims to evaluate the effectiveness of different exercise methods in improving health outcomes for postmenopausal women. As women go through menopause, they may experience changes such as decreased bone density, muscle weakness, and an increased risk of chronic diseases. Exercise is known to be beneficial in reducing these risks, but the best approach remains unclear.

In this clinical trial, participants will engage in structured exercise programs designed to improve bone health, strength, and overall well-being. The study will compare different types of exercises to determine which method provides the most benefits. By participating in this research, postmenopausal women can contribute to a better understanding of how exercise can enhance health during this stage of life.

This study is safe, and all exercises are guided by professionals. The results will help healthcare providers recommend the most effective exercise strategies for postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Being between 40-65 years of age Having a Body Mass Index (BMI) below 40 Scoring 68 or above on the System Usability Scale Having no orthopedic problems Completing the informed consent form Being within 5 years after a 12-month amenorrhea history

Exclusion Criteria:

* Presence of visual impairments Presence of musculoskeletal system disorders Presence of cognitive impairments Presence of joint range of motion limitations Presence of severe cardiac problems Participation in another program

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 12 months of amenore
Enrollment: 60 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Body Composition (Fat Mass, Lean Mass, and BMI) Assessed by Bioelectrical Impedance Analysis (BIA) | Baseline and Week 8
  Body composition (fat mass, lean mass, and BMI) measured using bioelectrical impedance analysis (BIA). Higher fat mass may be associated with lower exercise capacity.

SECONDARY OUTCOMES:
Menopause Symptom Assessment Scale Score | Baseline and Week 8
  Change in menopause symptoms assessed by the Menopause Symptom Assessment Scale. The scale consists of 11 items rated from 0 to 4, with a maximum score of 44. Higher scores indicate worse quality of life.
Fatigue Severity Scale Score | Baseline and Week 8
  Fatigue levels measured using the Fatigue Severity Scale (FSS), which consists of 9 questions scored between 0 and 7. A total score of 28 or above indicates severe fatigue.
Beck Depression Inventory (BDI) Score | Baseline and Week 8
  Depression levels assessed using the Beck Depression Inventory (BDI), with scores categorized into minimal, mild, moderate, and severe depression. A score above 30 indicates severe depression.
Pittsburgh Sleep Quality Index (PSQI) Score | Baseline and Week 8
  Sleep quality measured using the Pittsburgh Sleep Quality Index (PSQI), with a total score range of 0-21. A total score greater than 5 indicates poor sleep quality.
Short Form-36 (SF-36) Quality of Life Scale Score | Baseline and Week 8
  Quality of life will be measured using the Short Form-36 (SF-36) questionnaire, which evaluates physical and emotional well-being across 8 domains.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No